CLINICAL TRIAL: NCT00822354
Title: Tadalafil for the Treatment of Secondary Raynaud's Phenomenon
Brief Title: Tadalafil for the Treatment of Raynaud's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Anne Laumann, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU1199
Record Dates: First submitted 2008-05-31; First posted 2009-01-14 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Raynaud
Keywords: Secondary Raynaud's Phenomenon
MeSH Terms: conditions — Raynaud Disease | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects will receive tadalafil 20mg every other day for the first month, and then placebo for the second month.
  Interventions: Drug: Tadalafil
- 2 (Experimental): Subjects will receive placebo for the first month, and tadalafil 20mg orally every other day for the second month.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Subjects will be randomized to receive either tadalafil for the first month followed by placebo or placebo for the first month and followed by tadalafil
  Other Names: Cialis

SUMMARY:
The investigators propose that tadalafil will increase digital blood flow and improve the symptoms and signs of secondary Raynaud's phenomenon.

DETAILED DESCRIPTION:
The primary goal of our study is to decrease the frequency, duration and severity of vasospastic attacks in patients with secondary Raynaud's. The secondary goal is to document increased blood flow and lessened capillary dysfunction in these patients. Both of these goals are to be achieved using a course of treatment with Tadalafil.We anticipate a decrease in the frequency, duration and severity of Raynaud's attacks. Improved digital blood flow and digital blood pressures, and a decrease in digital capillary dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* active Raynaud's Phenomenon
* stable disease and medication requirements over the previous 2 months
* subjects willing and able to participate in study assessments
* ability to understand and sign informed consent
* ages 18 to 65, both sexes
* a diagnosis of diffuse or limited cutaneous sclerosis, MCTD using the American College Rheumatology criteria

Exclusion Criteria:

* uncontrolled HTN, DM, unstable disease, angina or using oral nitrates
* smoking, active alcoholism, drug abuse within 5 years
* abnormal renal function
* ulnar arterial occlusive disease as shown by a positive Allen Test
* Pregnant or breast feeding or considering preg. in next 4 months
* past or present major psych. illness
* allergy or sensitivity to tadalafil
* subject unable to understand protocol or give informed consent
* part. in another study trial within 30 days
* taking sildenafil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laumann, MBChB, MRCP, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Maltez N, Maxwell LJ, Rirash F, Tanjong Ghogomu E, Harding SE, Tingey PC, Wells GA, Tugwell P, Pope J. Phosphodiesterase 5 inhibitors (PDE5i) for the treatment of Raynaud's phenomenon. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD014089. doi: 10.1002/14651858.CD014089. PMID 37929840

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil Followed by Placebo: Subjects received tadalafil 20 mg every other day for four weeks followed by placebo every other day for four weeks. A one week washout occurred between the treatment and placebo periods.
- Placebo Followed by Tadalafil: Subjects received placebo every other day for four weeks, followed by tadalafil 20 mg every other day for four weeks. A one week washout occurred between the placebo and treatment periods.
Period: First Intervention (28 Days)
Arm/Group | Tadalafil Followed by Placebo | Placebo Followed by Tadalafil
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Period: Washout (7 Days)
Arm/Group | Tadalafil Followed by Placebo | Placebo Followed by Tadalafil
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention (28 Days)
Arm/Group | Tadalafil Followed by Placebo | Placebo Followed by Tadalafil
Started | 4 | 5
Completed | 3 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil Followed by Placebo | Placebo Followed by Tadalafil | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Raynaud's Phenomenon Attacks Per Day
Description: Subjects kept a daily record of the number of Raynaud's phenomenon attacks they experienced per day. Results are reported from data collected at Baseline/Week 0, Week 4, Week 5, and Week 9 visits. In subjects receiving tadalafil followed by placebo: Baseline/Week 0 data is Pre-treatment, Week 4 data corresponds to Week 4 of treatment, Week 5 data is Pre-placebo, and Week 9 data corresponds to Week 4 of placebo. In subjects receiving placebo followed by tadalafil: Baseline/Week 0 data is Pre-placebo, Week 4 data corresponds to Week 4 of placebo, Week 5 data is Pre-treatment, and Week 9 data corresponds to Week 4 of treatment.
Time Frame: 9 weeks
Population: Two of the ten enrolled subjects were excluded from analysis: one subject due to early withdrawal, and a second subject to avoid bias due to bilateral subclavian stent placement midway through the study. For subject 2, Week 5 data was used for both Pre-treatment and Pre-placebo because Baseline/Week 0 visit data was not obtained.
Measure: Median (Full Range); unit: Raynaud's attacks per day
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
Raynaud's attacks per day | 2.4 [0.2 to 8.1] | 1.1 [0.1 to 6.8] | 2.0 [0.3 to 6.7] | 2.3 [0.5 to 6.6]

2. Primary Outcome: Duration of Raynaud's Phenomenon Attacks
Description: Subjects kept a daily record of the number of Raynaud's phenomenon attacks they experienced per day and the duration of each attack. Results are reported from data collected at Baseline/Week 0, Week 4, Week 5, and Week 9 visits. In subjects receiving tadalafil followed by placebo: Baseline/Week 0 data is Pre-treatment, Week 4 data corresponds to Week 4 of treatment, Week 5 data is Pre-placebo, and Week 9 data corresponds to Week 4 of placebo. In subjects receiving placebo followed by tadalafil: Baseline/Week 0 data is Pre-placebo, Week 4 data corresponds to Week 4 of placebo, Week 5 data is Pre-treatment, and Week 9 data corresponds to Week 4 of treatment.
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
minutes | 5.7 [0.1 to 60.4] | 11.4 [1 to 35.4] | 1.2 [.1 to 13.2] | 14.2 [5.6 to 39.5]

3. Primary Outcome: Raynaud Severity Visual Analog Score (VAS)
Description: The VAS is a 100 millimeter (mm) line where 0 mm (left boundary) represents Raynaud's disease of low severity, and 100 mm (right boundary) represents extremely severe Raynaud's disease. The subject makes a vertical mark on the VAS to indicate the severity of Raynaud's disease over the past two weeks. The Raynaud's severity score is the distance from the left boundary to the vertical mark in mm. Results are reported from data collected at Baseline/Week 0, Week 4, Week 5, and Week 9 visits. In subjects receiving tadalafil followed by placebo: Baseline/Week 0 data is Pre-treatment, Week 4 data corresponds to Week 4 of treatment, Week 5 data is Pre-placebo, and Week 9 data corresponds to Week 4 of placebo. In subjects receiving placebo followed by tadalafil: Baseline/Week 0 data is Pre-placebo, Week 4 data corresponds to Week 4 of placebo, Week 5 data is Pre-treatment, and Week 9 data corresponds to Week 4 of treatment.
Time Frame: 9 weeks
Population: Two of the ten enrolled subjects were excluded from analysis: one subject due to early withdrawal, and a second subject to avoid bias due to bilateral subclavian stent placement midway through the study.
Measure: Median (Full Range); unit: millimeters
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
millimeters | 39 [19 to 100] | 16.5 [1 to 55] | 51.5 [11 to 71] | 37 [9 to 69]

4. Secondary Outcome: Digital Blood Pressure
Description: Results are reported from data collected at Baseline/Week 0, Week 4, Week 5, and Week 9 visits. In subjects receiving tadalafil followed by placebo: Baseline/Week 0 data is Pre-treatment, Week 4 data corresponds to Week 4 of treatment, Week 5 data is Pre-placebo, and Week 9 data corresponds to Week 4 of placebo. In subjects receiving placebo followed by tadalafil: Baseline/Week 0 data is Pre-placebo, Week 4 data corresponds to Week 4 of placebo, Week 5 data is Pre-treatment, and Week 9 data corresponds to Week 4 of treatment.
Time Frame: 9 weeks
Population: Two of the ten enrolled subjects were excluded from analysis: one subject due to early withdrawal, and a second subject to avoid bias due to bilateral subclavian stent placement midway through the study. For subject 10, Week 2 data was used for Week 4 of placebo because digital blood pressure data was not obtained at the Week 4 visit.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
mm Hg | 97 [44 to 127] | 80 [60 to 127] | 84 [71 to 121] | 80 [67 to 121]

5. Secondary Outcome: Capillary Diameter
Description: as for outcome 4
Time Frame: 9 weeks
Population: Two of the ten enrolled subjects were excluded from analysis: one subject due to early withdrawal, and a second subject to avoid bias due to bilateral subclavian stent placement midway through the study. For subject 8, Baseline/Week 0 data was used for both Pre-treatment and Pre-placebo, and Week 2 data was used for Week 4 of placebo.
Measure: Median (Full Range); unit: micrometers
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
micrometers | 9.3 [6.5 to 19.3] | 10 [3.6 to 19.3] | 10.7 [5.7 to 25.7] | 10 [7.9 to 17.1]

6. Primary Outcome: Raynaud's Condition Score (RCS) Visual Analog Scale (VAS)
Description: The VAS is a 100 millimeter (mm) line where 0 mm (left boundary) represents no difficulty with Raynaud's disease, and 100 mm (right boundary) represents extreme difficulty with Raynaud's disease. The subject makes a vertical mark on the VAS to indicate difficulty experienced that day with Raynaud's disease. The RCS is the distance from the left boundary to the vertical mark in mm. Results are reported from data collected at Baseline/Week 0, Week 4, Week 5, and Week 9 visits. In subjects receiving tadalafil followed by placebo: Baseline/Week 0 data is Pre-treatment, Week 4 data corresponds to Week 4 of treatment, Week 5 data is Pre-placebo, and Week 9 data corresponds to Week 4 of placebo. In subjects receiving placebo followed by tadalafil: Baseline/Week 0 data is Pre-placebo, Week 4 data corresponds to Week 4 of placebo, Week 5 data is Pre-treatment, and Week 9 data corresponds to Week 4 of treatment.
Time Frame: 9 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: millimeters
Arm/Group | Pre-treatment | Week 4 of Treatment | Pre-placebo | Week 4 of Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
millimeters | 38.5 [7 to 84] | 9 [0 to 57] | 35 [0 to 60] | 26 [0 to 70]

ADVERSE EVENTS:
Groups:
- Tadalafil: Subjects received tadalafil 20 mg every other day for four weeks.
- Placebo: Subjects received placebo every other day for four weeks
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes